CLINICAL TRIAL: NCT00830934
Title: Randomised Controlled Trial for the Treatment of Pelvic Girdle Pain in Pregnancy
Brief Title: Trial for the Treatment of Pelvic and Back Pain in Pregnancy
Acronym: GRIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University College Cork (Other)
Responsible Party: Professor Richard A Greene, Cork University Maternity Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GRIP1
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Pelvic Girdle Pain; Symphysio Pubic Dysfunction
Keywords: pelvic girdle pain; symphysio pubic dysfunction; group care; individual care
MeSH Terms: conditions — Pelvic Girdle Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Individual care (Active Comparator): The first treatment group (individual care group) will involve 3 sessions held weekly. Each session will last approximately 45 minutes.
  Interventions: Procedure: Individual care
- Group care (Experimental): The second treatment group (group care group) will be assigned to weekly group exercise classes, focusing on core stability and strengthening exercises. Classes will last one hour and will be conducted for 4 weeks. In both treatment groups pain scores will be followed up for 1 week post last treatment.
  Interventions: Procedure: group care

INTERVENTIONS:
Procedure: Individual care — The first treatment group (individual care group) will involve 3 sessions held weekly. Each session will last approximately 45 minutes.
  Arms: Individual care
Procedure: group care — The second treatment group (group care group) will be assigned to weekly group exercise classes, focusing on core stability and strengthening exercises. Classes will last one hour and will be conducted for 4 weeks. In both treatment groups pain scores will be followed up for 1 week post last treatment.
  Arms: Group care

SUMMARY:
The investigators aim to conduct a prospective open label randomized controlled trial to test the hypothesis that following initial assessment by a physiotherapist, group care exercise class is as effective in reducing pain as individual physiotherapy care.

DETAILED DESCRIPTION:
Back pain is reported to affect at least 75% of women at some stage during their pregnancy. In the United States one review found that approximately a third of women find back pain in pregnancy a severe problem. It has been reported that 20% of all pregnant women suffer from the condition to such an extent that they require medical help. Six years after pregnancy, problems remain in about 7% of women with PGP, causing severe disability and reducing ability to work. The increase in back pain in pregnancy occurs most likely as a result of the natural underlying posture deviations been accentuated in pregnancy. Anterior displacement of the sacrum, posterior displacement of the trunk and a significant increase in the anterior tilt of the pelvis results in exaggerated lordosis of the lower back.

Stretching, weakness, and separation of abdominal muscles further impede neutral posture and place even more strain on paraspinal muscles. Joint laxity in the anterior and posterior longitudinal ligaments of the lumbar spine puts strain on the lumbar spine and there is widening and increased mobility of the sacroiliac joints and pubic symphysis to facilitate the baby's passage through the birth canal.

A significant cause of back pain in pregnancy appears to result from pelvic girdle pain (PGP). Back pain in pregnancy is more common in women with pre-existing back pain, back pain in a previous pregnancy, advanced maternal age and multiparity. Despite the high incidence of back pain in pregnancy (75% of women attending antenatal clinics at Cork University Maternity Hospital) only a fraction of women (25% in the same audit) report back pain to their health care providers presumably due to their perception that there are minimal interventions for the safe treatment of back pain in pregnancy. Similar results have been shown in other studies.

A Cochrane review on interventions for preventing and treating pelvic and back pain in pregnancy republished in October 2008 found no studies dealing specifically with prevention of back or pelvic pain in pregnancy. They included eight studies (1305 participants) that examined the effects of adding various pregnancy-specific exercises, physiotherapy, acupuncture and pillows compared with usual prenatal care. They concluded that all but one study had moderate to high potential for bias. Adding pregnancy specific exercises, physiotherapy or acupuncture to usual prenatal care appears to relieve back or pelvic pain more than usual prenatal care alone, although the effects appear small. Recent trials investigating the effect of acupuncture on PGP concluded that acupuncture and stabilising exercises constitute efficient complements to standard treatment for the management of PGP in pregnancy but acupuncture alone has no significant effect on pain or on the degree of sick leave compared with non penetrating sham acupuncture.

The pain of PGP is experienced between the posterior iliac crest and the gluteal fold, particularly in the vicinity of the sacroiliac joints. The endurance capacity for standing, walking and sitting is diminished. Diagnosis can only be reached after exclusion of lumbar causes and this diagnosis should be based on a medical history, a physical standardised examination with specific clinical tests that reproduce pain in the pelvic girdle.

The European guidelines state that available evidence is insufficient to recommend any particular treatment modality.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (primigravida and multigravida) from 20-35 weeks of gestation attending Cork University Maternity Hospital (CUMH) low risk antenatal clinics who are referred to the physiotherapy department by their health care provider or following self referral with back pain or pelvic pain will be assessed for inclusion in the trial.
* Women referred to the physiotherapy department with symptoms of PGP will be assessed on presentation by a one of six departmental physiotherapists specializing in women's health.
* To make the diagnosis of PGP the following tests will be performed as per the European Guidelines on the diagnosis and treatment of Pelvic Girdle Pain and a pain history taken as detailed.
* Sacroiliac joint assessment

  1. Posterior pelvic pain provocation test (P4)
  2. Gaenslen´s test.
  3. Compression of ASIS
  4. Distraction SIJ pain provocation test
  5. Assessment of Sulci depth in lumbar spine in neutral and extension
* Functional pelvic test 6.Active straight leg raise test (ASLR).
* Pain history (according to the criteria of Ostgaard)

  7.It is recommended that a pain history be taken with specific attention paid to pain patterns and irritability of PGP.

  8.There must be no nerve root syndrome. 9.The severity of pain must be related to motion.
* The diagnosis of PGP will be made if the patient has 2 or more of criteria 1-4 (Laslett's criteria) in combination with a negative McKenzie and negative neurological examination. Criteria 5-9 will be performed and assessed to try and improve diagnostic sensitivity and specificity as well as help exclude other pathologies that may cause pelvic and back pain.

Exclusion Criteria:

1. Women with other pain conditions, history of orthopaedic disease or surgery in the spine or pelvic girdle systemic disorders or if attending the high risk antenatal clinic in CUMH will be excluded from the study.
2. If women volunteered a history of sexual abuse at any point of the study they would be excluded from the trial.
3. Women who do not speak English fluently.
4. Women with non viable pregnancies.
5. Women who have already received treatment for PGP outside of this trial.
6. Pregnant women who present who will not be booking at CUMH for their pregnancy or are not resident in the South West of Ireland
7. Women with a history of severe PGP in previous pregnancies. Severe PGP will be defined as occurring less than 20 weeks gestation in a previous pregnancy or requiring crutches in a previous pregnancy or women with a history of PGP in 2 or more previous pregnancies.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2009-04; Primary Completion 2010-03 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
A reduction in the current intensity of PGP related to motion on a 100-point Visual analogue score (VAS). | VAS recorded twice daily every morning and evening by the patient beginning at initial assessement (week one) and continuing until 1 week following the course of treatment. (week 5 for individual care group and week 6 for group treatment group)

SECONDARY OUTCOMES:
Admission to hospital with PGP | From initial assessment and diagnosis until delivery.
Frequency of sick leave from work due to PGP | From initial assessment and diagnosis to delivery.
Representation at the physiotherapy department during the trial period. | While receiving treatment which the patient has been randomized to.(from week 1 to week 5 for individual care group and week 6 for group treatment group)
Representation at the physiotherapy department | After the trial treatment period prior to delivery. (week 5 for individual care group and week 6 for group treatment group)
Number of patients requiring the combination of crutches and Tubigrip ® (elasticated tubular support bandage). | During the antenatal period.
Number of patients induced or delivered earlier than their estimated date of delivery due to severe PGP. | During course of current pregnancy
Patient satisfaction measured via the CSQ-18B | Following the third treatment session i.e. 4 weeks following initial assessment and randomization.
Patient specific functional scale (PSFS). | This will be measured at initial assessment and following the third treatment i.e. 4 weeks following initial assessment and randomization.
Active straight leg raise. | This will be measured at initial assessment and following the third treatment i.e. 4 weeks following initial assessment and randomization.
Gestational age at delivery | During current pregnancy
Birthweight at delivery. | During current pregnancy
Mode of delivery: Either normal vaginal delivery, instrumental delivery or caesarean section. | During current pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Maternity Hospital, Cork, Cork, Ireland

REFERENCES:
- [Background] Kristiansson P, Svardsudd K, von Schoultz B. Back pain during pregnancy: a prospective study. Spine (Phila Pa 1976). 1996 Mar 15;21(6):702-9. doi: 10.1097/00007632-199603150-00008. PMID 8882692
- [Background] Ostgaard HC, Zetherstrom G, Roos-Hansson E. Back pain in relation to pregnancy: a 6-year follow-up. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2945-50. doi: 10.1097/00007632-199712150-00018. PMID 9431631
- [Background] Foti T, Davids JR, Bagley A. A biomechanical analysis of gait during pregnancy. J Bone Joint Surg Am. 2000 May;82(5):625-32. PMID 10819273
- [Background] Gilleard W, Crosbie J, Smith R. Effect of pregnancy on trunk range of motion when sitting and standing. Acta Obstet Gynecol Scand. 2002 Nov;81(11):1011-20. doi: 10.1034/j.1600-0412.2002.811104.x. PMID 12421168
- [Background] Marnach ML, Ramin KD, Ramsey PS, Song SW, Stensland JJ, An KN. Characterization of the relationship between joint laxity and maternal hormones in pregnancy. Obstet Gynecol. 2003 Feb;101(2):331-5. doi: 10.1016/s0029-7844(02)02447-x. PMID 12576258
- [Background] Pennick VE, Young G. Interventions for preventing and treating pelvic and back pain in pregnancy. Cochrane Database Syst Rev. 2007 Apr 18;(2):CD001139. doi: 10.1002/14651858.CD001139.pub2. PMID 17443503
- [Background] Elden H, Fagevik-Olsen M, Ostgaard HC, Stener-Victorin E, Hagberg H. Acupuncture as an adjunct to standard treatment for pelvic girdle pain in pregnant women: randomised double-blinded controlled trial comparing acupuncture with non-penetrating sham acupuncture. BJOG. 2008 Dec;115(13):1655-68. doi: 10.1111/j.1471-0528.2008.01904.x. Epub 2008 Oct 15. PMID 18947338
- [Background] Elden H, Ladfors L, Olsen MF, Ostgaard HC, Hagberg H. Effects of acupuncture and stabilising exercises as adjunct to standard treatment in pregnant women with pelvic girdle pain: randomised single blind controlled trial. BMJ. 2005 Apr 2;330(7494):761. doi: 10.1136/bmj.38397.507014.E0. Epub 2005 Mar 18. PMID 15778231
- [Background] Vleeming A, Albert HB, Ostgaard HC, Sturesson B, Stuge B. European guidelines for the diagnosis and treatment of pelvic girdle pain. Eur Spine J. 2008 Jun;17(6):794-819. doi: 10.1007/s00586-008-0602-4. Epub 2008 Feb 8. PMID 18259783
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Stratford, P., Gill, C., Westaway, M., & Binkley, J., Assessing disability and change on individual patients: a report of a patient specific measure. Physiotherapy Canada, 47, 258-263. 1995
- [Background] Leadbetter RE, Mawer D, Lindow SW. The development of a scoring system for symphysis pubis dysfunction. J Obstet Gynaecol. 2006 Jan;26(1):20-3. doi: 10.1080/01443610500363915. PMID 16390703
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Kelly AM. Does the clinically significant difference in visual analog scale pain scores vary with gender, age, or cause of pain? Acad Emerg Med. 1998 Nov;5(11):1086-90. doi: 10.1111/j.1553-2712.1998.tb02667.x. PMID 9835471
- [Background] Ostgaard HC, Zetherstrom G, Roos-Hansson E, Svanberg B. Reduction of back and posterior pelvic pain in pregnancy. Spine (Phila Pa 1976). 1994 Apr 15;19(8):894-900. doi: 10.1097/00007632-199404150-00005. PMID 8009346
- [Background] Laslett M, Young SB, Aprill CN, McDonald B. Diagnosing painful sacroiliac joints: A validity study of a McKenzie evaluation and sacroiliac provocation tests. Aust J Physiother. 2003;49(2):89-97. doi: 10.1016/s0004-9514(14)60125-2. PMID 12775204
- [Background] Altman DG, Schulz KF, Moher D, Egger M, Davidoff F, Elbourne D, Gotzsche PC, Lang T; CONSORT GROUP (Consolidated Standards of Reporting Trials). The revised CONSORT statement for reporting randomized trials: explanation and elaboration. Ann Intern Med. 2001 Apr 17;134(8):663-94. doi: 10.7326/0003-4819-134-8-200104170-00012. PMID 11304107
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066